CLINICAL TRIAL: NCT04153968
Title: Determination of Relative Bioavailability, Bioconversion and Bioefficacy of β-cryptoxanthin in Comparison to β-carotene From Biofortified Maize and External Stable Isotopes Using Compartmental Modelling
Brief Title: Bioefficacy of Beta-cryptoxanthin From Biofortified Maize
Acronym: BIOCRYPT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Newcastle University (Other)
Collaborators: International Food Policy Research Institute (Other); Penn State University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: BH183438
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Vitamin A Deficiency
MeSH Terms: conditions — Vitamin A Deficiency | interventions — retinol acetate

STUDY DESIGN:
Intervention Model Description: The study is designed in two phases to allow the research team to firstly determine the absorption and bioconversion kinetics of pure βCX and provide external validation for single-sample prediction methods. The second phase aims to test the bioavailability of both pVACs in maize by comparing a high βCX:βC variety to a low βCX:βC variety in combination with external [13C]-labelled pVACs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1 (Experimental): Determination absorption and bioconversion kinetics of [13C14]β-cryptoxanthin and provide external validation for single-sample prediction methods.
  Interventions: Dietary Supplement: β-cryptoxanthin
- Phase 2 (Experimental): Test the bioefficacy of provitamin A carotenoids (pVACs) in maize by comparing a high β-cryptoxanthin:β-carotene (βCX:βC) variety to a low βCX:βC variety in combination with external [13C]-labelled pVACs.
  Interventions: Dietary Supplement: β-cryptoxanthin

INTERVENTIONS:
Dietary Supplement: β-cryptoxanthin — Phase 1:
  2.0mg of [13C14]β-cryptoxanthin, 1.0mg of [13C10]β-carotene and 0.4mg [2H6]retinyl acetate are given in sunflower oil at Time 0.
  Phase 2:
  1.5mg of [13C14]β-cryptoxanthin, 0.75mg of [13C10]β-carotene, 0.4mg [2H6]retinyl acetate are given in sunflower oil along with 0.25mg β-carotene and 0.5mg β-cryptoxanthin from maize are given at Time 0.
  Then, 0.75mg of [13C14]β-cryptoxanthin, 1.5mg of [13C10]β-carotene, and 0.4mg [2H6]retinyl acetate are given in sunflower oil along with 0.5mg β-carotene and 0.25mg β-cryptoxanthin from maize are given on day 21.
  Other Names: β-carotene; retinyl acetate

SUMMARY:
Since no quantitative information currently exists on how effectively the pro-vitamin A carotenoid (pVAC) β-cryptoxanthin (βCX) is converted to vitamin A (VA) in humans, this proof of principle study aims to compare the efficacy of both βCX and β-carotene (βC) to yield VA from biofortified maize. This data is critical before the breeding strategy for biofortified maize is directed towards high βCX-containing varieties in order to reduce VA deficiency in low-income countries.

DETAILED DESCRIPTION:
Despite advances in reducing vitamin A (VA) deficiency worldwide, the prevalence remains highest and unchanged in sub-Saharan Africa and South Asia. Efficacy studies have demonstrated that increasing provitamin A carotenoid (pVAC) intake through consuming pVAC biofortified crops results in increased circulating β-carotene (βC) and VA body stores. It has also been shown that consumption of biofortified maize improved VA total body stores (TBS) as effectively as preformed VA supplementation, and significantly improved visual function in marginally VA deficient children. Despite the fact that βC is the primary focus of breeding programs for pVAC biofortified maize, there is convincing evidence that comparable dietary intakes of βC and β-cryptoxanthin (βCX) would result in 7-fold greater concentrations of βCX in blood.

The study is designed to determine for the first time the bioefficacy of βCX in comparison to βC in humans using state of the art isotope dilution techniques in combination with compartmental modelling. The project is conducted in two phases: Phase 1) the determination of best time points for assessment of βCX bioconversion, intestinal and postintestinal bioefficacy as well as quantifying TBS of VA in healthy volunteers; Phase 2) to test the bioefficacy of βCX and βC in maize by comparing a high βCX and low βC maize variety to a high βC and low βCX maize variety.

Phase 1 of the study involves 1 long study day (D0), where 10 ml of blood will be taken every 2 hours, via cannulation, for a total of 12 hours (70 ml of blood total). Subsequently, there are 13 followup visits on the mornings of Days 1, 2, 4, 7, 11, 14, 21, 28, 35, 49, 63, 77, and 91 where one 10 ml blood sample is taken.

Phase 2 of the study involves 2 whole days (D0 and D21) where approximately 10 ml of blood will be taken every 30-60 minutes, via cannulation, for a total of 8 hours (110 ml of blood total). Subsequently, there are 3 follow-up visits on the mornings of Days 1, 7, and 22 where one 10 ml blood sample is taken on each occasion.

In the mornings of the long/whole study days at either D0 or D21, participants will receive the muffin test meal before stable isotopes, dissolved in sunflower oil, are administered via oral pipette. At D0 or D21, the total dose of pVACs (labelled and unlabelled carotenoids) consumed in the muffin and oil is 3 mg alongside 0.4 mg of pre-formed VA.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Females who are pregnant or lactating.
* Not disclosing use and type of contraceptives.
* Acute or chronic illness.
* Concurrent participation in another study.
* Unwillingness to discontinue personal nutritional supplements/vitamins.
* Major food allergies/intolerance to study ingredients.
* Previous history of anorexia or bulimia.
* Inability to refrain from drinking alcohol when requested.
* Fat mal-absorptive disorders or iron deficiency anaemia.
* Dietary preformed vitamin A intake >600 µg/d.
* BMI <20 and >29 kg/m2.
* Smoking.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Bioefficacy of β-cryptoxanthin | Phase 1 = 91 days. Phase 2 = 22 days.
  Plasma concentrations of [13C14]-β-cryptoxanthin, [13C7]-retinyl esters, and [13C7]-retinol.

CONTACTS AND LOCATIONS:
Locations (1):
- Newcastle University, Newcastle upon Tyne, Tyne & Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No